CLINICAL TRIAL: NCT02143583
Title: Long-term Follow-up of a Multicentre, Randomized, Double-blind, Placebo-controlled Trial (AN004T) Assessing the Efficacy and Tolerability of 2 Dosing Regimens of AllerT in Adult Subjects Allergic to Birch Pollen
Brief Title: Follow-up of Study AN004T to Assess the Persistence of AllerT Efficacy During the 2nd to 4th Season After Treatment
Status: Completed | Type: Observational
Sponsor: Anergis (Industry)
Responsible Party: Sponsor
Other Study IDs: AN005T; 2013-003881-15 (EudraCT Number)
Record Dates: First submitted 2014-05-02; First posted 2014-05-21 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Birch Pollen Allergy
Keywords: rhinoconjunctivitis; birch pollen; desensitization; allergen immunotherapy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AllerT 100 μg: patients having received AllerT at a first dose of 50 μg and 4 maintenance doses of 100 μg in study AN004T
- AllerT 50 μg: patients having received AllerT at a first dose of 25 μg and 4 maintenance doses of 50 μg in study AN004T
- Placebo: Patients having received Placebo (i.e., adjuvant alone) delivered in the same manner as AllerT in study AN004T

SUMMARY:
Study aiming to evaluate the efficacy of a 2-month pre-seasonal treatment with an AllerT 50 µg or 100 µg maintenance dose administered in previous study AN004T in reducing symptoms of allergic rhinoconjunctivitis during the 2nd following birch pollen season.

DETAILED DESCRIPTION:
Multicenter, international, parallel-group follow-up study of subjects randomized and treated in Study AN004T (AllerT 100 µg, AllerT 50 µg, placebo) and followed over the 2nd, and if appropriate, the 3rd and 4th birch pollen seasons in this study (still double-blind during the 1st year, open-label in the 2nd and 3rd years).

ELIGIBILITY:
Inclusion Criteria:

1. Any subject having been randomized in the AN004T trial and had received at least one injection
2. Any subject having been informed and provided signed consent for participating in the trial and willing to follow all planned trial assessments

Exclusion Criteria:

1. Any subject having received specific immunotherapy against birch pollen or a tree pollen mix including birch pollen at any time since AN004T and before Visit 1
2. Any subject intending to travel during the birch pollen season outside of the birch pollination area for more than 7 consecutive days
3. Any subject unable or unwilling to record allergy symptoms and medications daily during the following birch pollen season using an electronic diary device
4. Any subject not covered by medical insurance
5. Any subject having received immunosuppressive medication within 4 weeks prior to inclusion, or planned to be used during the trial period
6. Any subject having received systemic or local antihistamines, oral or inhaled corticosteroids or under anti depressant medication with antihistamine effect within 2 weeks prior to inclusion
7. Any subject having used any investigational or non-registered drug, vaccine, or medical device within 4 weeks prior to inclusion, or planned to use such treatments during the trial period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects with moderate to severe allergic rhiniconjunctivitis to birch pollen
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Framçois SPERTINI, MD, Principal Investigator — University of Lausanne Hospitals
Locations (22):
- Denmark (3):
  - Allergiklinikken, Hellerup, Copenhagen
  - Lungemedicinsk Forskningsafdeling, Aarhus
  - Klinisk Institute, Odense
- Hopitaux Universitaires de Strasbourg, Strasbourg, France
- Latvia (2):
  - Viktorija Vevere private practice of Allergology, Rēzekne
  - Center of examination and treatment of allergic diseases, Riga
- Lithuania (4):
  - Kaunas Clinics University Hospital, Kaunas
  - Allergy Clinic JSC Perspektyvos, Vilnius
  - Vilnius University Hospital, Vilnius
  - Antakalnio affiliation of the Vilnius City Allergy Center, Vilnius
- Poland (8):
  - SPZOZ Uniwersytecki Szpital Kliniczny - Allergology, Lodz
  - Alergologii Centrum, Lodz
  - Alergotest, Lublin
  - Alergo-Med, Tarnów
  - Centrum Alergologii IRMED, Warsaw
  - Silesian Piasts University of Medicine in Wrocław, Wroclaw
  - Aler-med, Wroclaw
  - NZOZ Przychodnia Lekarska Hipokrates, Zabrze
- Sweden (3):
  - University hospital Skane, Lund
  - Orebro University Hospital, Örebro
  - Lungavdelningen, Vastmanlands, Västerås
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AllerT 100 μg | AllerT 50 μg | Placebo
Started | 62 | 66 | 68
Completed | 61 | 66 | 66
Not Completed | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — husband illness | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set : subjects having received at least one injection of AllerT or placebo in AN004T and successfully screened in AN005T
Groups:
- Total: Total of all reporting groups
Arm/Group | AllerT 100 μg | AllerT 50 μg | Placebo | Total
Number analyzed (Participants) | 62 | 66 | 68 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (9.0) | 37.9 (9.4) | 35.5 (9.3) | 37.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 37 | 34 | 101
  Male | 32 | 29 | 34 | 95

OUTCOME MEASURES:

1. Primary Outcome: Average of the Combined Rhinoconjunctivitis Symptom and Medication Score (RSMS) Obtained Daily During the Birch Pollen Season
Description: The scale range is from 0 to 3. Lower is the the RSMS value, better is the efficacy as this implies that lower is the symptoms and concomitant medication intake by the patient The RSMS includes 2 subscales : the Rhinoconjunctivitis Symptom Score (RSS) with a range of values from 0 to 3 and the Rhinoconjunctivitis Medication Score Score (RMS) with also a range of values from 0 to 3 The RSMS is the sum of the RSS and RMS divided by 2 The Rhinoconjunctivitis Symptom Score (RSS) comprises 6 different symptoms from the nose and eyes. The sum of the 6 symptom scores divided by 6 will be used as the RSS (scale of 0 to 3).
  The daily Rhinoconjunctivitis Medication Score (RMS) will be determined by assigning daily scores as follows:
  0 = no medication
  1. = subject took topical antihistamine
  2. = subject took oral antihistamine
  3. = subject took oral corticosteroids
Time Frame: from the first of 3 consecutive days with a regional pollen count > 10 grains/m3 to the earliest between the 42nd day after the start of the season and the last day in the last occurrence of 3 consecutive days with a regional pollen count ≥ 10 grains/m3
Population: Modified-ITT analysis set : participants having received at least 4 injections of AllerT or placebo in AN004T
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AllerT 100 μg | AllerT 50 μg | Placebo
Number analyzed (Participants) | 57 | 64 | 68
units on a scale | 0.853 (0.524) | 0.795 (0.421) | 0.959 (0.487)

2. Secondary Outcome: Average of the Total Score of the Validated Mini Rhinoconjunctivitis Quality-of-life Questionnaire© (Mini RQLQ) Obtained Weekly During the Birch Pollen Season
Description: The Mini-RQLQ will be used. This evaluation tool includes 14 questions assessing 5 domains (activity limitation, practical problems, nose symptoms, eye symptoms, and non-nose/eye symptoms).
  For each question the answer is quoted from 0: "no troubled" to 6: "extremely troubled"; then the average of the score for the 14 questions is calculated resulting in a scale from 0 to 6, 0 being the best case and 6 the worst case
Time Frame: between the 42nd day after the start of the season and the last day in the last occurrence of 3 consecutive days with a regional pollen count ≥ 10 grains/m3
Population: Modified-ITT analysis set : patients having received at least 4 injections of AllerT or placebo in AN004T
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AllerT 100 μg | AllerT 50 μg | Placebo
Number analyzed (Participants) | 57 | 64 | 68
units on a scale | 1.486 (1.017) | 1.479 (0.879) | 1.767 (1.054)

ADVERSE EVENTS:
Arm/Group | AllerT 100 μg | AllerT 50 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/62 | 2/66 | 0/68
Other Adverse Events (participants affected / at risk) | 2/62 | 1/66 | 4/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AllerT 100 μg (N=62) | AllerT 50 μg (N=66) | Placebo (N=68)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Non drug-related
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Non drug-related
Threatened labor (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Non drug-related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AllerT 100 μg (N=62) | AllerT 50 μg (N=66) | Placebo (N=68)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4) — Non drug-related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI coordinator of the study owns shares in Anergis SA